CLINICAL TRIAL: NCT04205318
Title: Impact of FTO Gene Variants and Lifestyle Factors on Obesity Traits in a Turkish Population
Brief Title: FTO Gene Variants and Diet in Obesity
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: University of Reading (Other); The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, ZEHRA BUYUKTUNCER, Professor, Hacettepe University
Other Study IDs: GO15/612-11
Record Dates: First submitted 2019-07-21; First posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-08

CONDITIONS: Obesity; Diet Habit; Genetic Predisposition
Keywords: obesity; gene-diet interaction; FTO gene variant
MeSH Terms: conditions — Obesity; Feeding Behavior; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study: obese (BMI ≥25.00 kg/m2, n=200)
- control: non-obese (BMI= 18.50-24.99 kg/m2, n=200)

SUMMARY:
Studies have shown that the effect of fat mass and obesity-associated (FTO) gene on obesity is modulated by lifestyle factors. Hence, we aimed to determine whether two single nucleotide polymorphisms (SNPs) in the FTO gene are associated with obesity and to assess whether these associations were modified by lifestyle factors. The study included 200 obese and 200 non-obese individuals from Turkey. Our study suggests that the effect of the SNPs on obesity traits is likely to be influenced by lifestyle factors in this Turkish population.

ELIGIBILITY:
Inclusion Criteria:

1. attending routine outpatient visits,
2. aged 24 to 50 years,
3. having a BMI ≥ 18.50 kg/m2

Ages: 24 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 400 unrelated individuals, aged 24-50 years
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Genetic analysis of two SNPs at FTO gene | up to 36 weeks
  FTO SNPs rs9939609 and rs10163409
Anthropometric measurements | up to 36 weeks
  Body mass index, waist circumference, hip circumference, body composition
Biochemical measurements | up to 36 weeks
  lipid profile, glucose, insulin, adiponectin

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Buyuktuncer, Principal Investigator — Hacettepe University, Department of Nutrition and Dietetics, Ankara, TURKEY; Vimales Karani Santhanakrishnan, Principal Investigator — Department of Food and Nutritional Sciences, University of Reading, UK
Locations (1):
- Zehra Buyuktuncer, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No